CLINICAL TRIAL: NCT00524459
Title: Phase II Study of Neoadjuvant Pegylated Liposomal Doxorubicin and Docetaxel in Locally Advanced Operable Breast Cancer
Brief Title: Pegylated Liposomal Doxorubicin and Docetaxel in Treating Women With Locally Advanced Breast Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by sponsor due to lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: I 75506; RPCI-I-75506
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel
Drug: pegylated liposomal doxorubicin hydrochloride
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal doxorubicin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving them before surgery may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving liposomal doxorubicin together with docetaxel before surgery and to see how well it works in treating women with locally advanced breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the rate of pathological complete response and clinical complete response in women with locally advanced breast cancer treated with pegylated doxorubicin hydrochloride liposome and docetaxel.

Secondary

* To assess the overall clinical local regional response in patients treated with this preoperative chemotherapy regimen.
* To evaluate the number of patients who would have required a mastectomy upfront but who underwent breast conservation therapy instead after neoadjuvant chemotherapy.
* To assess the safety, particularly with regard to neutropenia and cardiac toxicity, of pegylated doxorubicin hydrochloride liposome and docetaxel.

OUTLINE: This is a multicenter study.

Patients receive pegylated doxorubicin hydrochloride liposome IV over 90 minutes and docetaxel IV over 90 minutes on day 1. Patients receive pegylated filgrastim subcutaneously on days 2 or 3 post-chemotherapy in courses 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Within 8 weeks after completion of chemotherapy, patients undergo a lumpectomy or mastectomy to remove the tumor. Some patients may receive additional therapy after surgery, including hormonal therapy, chemotherapy, or radiotherapy.

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer using core biopsies

  * Locally advanced disease
  * Resectable disease
  * Fine needle aspiration cytology allowed and must demonstrate invasive adenocarcinoma
* No more than 8 weeks since initial cytologic or histologic diagnosis of breast cancer
* Tumor must meet the following criteria:

  * Palpable on clinical examination and confined to either the breast or to the breast and ipsilateral axilla
  * Measured clinically as greater than 2 cm in size (T2)
* Patients with skeletal pain are eligible if bone scan and/or roentgenological examination fail to disclose metastatic disease

  * Suspicious findings must be confirmed as benign by x-ray, MRI scan, or biopsy
* Hormonal status not specified

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Female
* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 10 years
* Platelet count ≥ 100,000/mm³
* ANC ≥ 1,500/mm³
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin normal
* AST or ALT normal
* Alkaline phosphatase normal
* Serum creatinine normal
* Negative pregnancy test
* Fertile patients must use effective contraception (e.g., abstinence, intrauterine device, barrier device with spermicide, or surgical sterilization) during and for 3 months after completion of study therapy
* Normal cardiac function by LVEF or MUGA scan
* Patients with prior non-breast malignancies are eligible if they have been disease-free for ≥ 10 years

  * The following are allowed even if diagnosed within the past 10 years:

    * Squamous or basal cell carcinoma of the skin that has been effectively treated
    * Carcinoma in situ of the cervix that has been treated by operation only
    * Lobular carcinoma in situ of the ipsilateral or contralateral breast treated by segmental resection only

Exclusion criteria:

* Pregnant or lactating women
* Male patients
* Hyperbilirubinemia
* Female patients with 1 or more of the following conditions:

  * Ulceration, erythema, infiltration of the skin (complete fixation), or peau d'orange (edema) of any magnitude

    * Tethering or dimpling of the skin or nipple inversion should not be interpreted as skin infiltration
  * Ipsilateral lymph nodes that are clinically fixed to one another or to other structures (N2 disease)
  * Bilateral malignancy or a mass in the opposite breast suspicious for malignancy, unless there is biopsy proof that the mass is not malignant
  * Suspicious palpable nodes in the contralateral axilla or palpable supraclavicular or infraclavicular nodes, unless there is biopsy evidence that these are not involved with the tumor
* Nonmalignant systemic disease (e.g., cardiovascular, renal, or hepatic) that would preclude study therapy
* Active cardiac disease that would preclude the use of doxorubicin hydrochloride, including any of the following:

  * Documented myocardial infarction
  * Angina pectoris that requires the use of antianginal medication
  * History of documented New York Heart Association class II-IV heart failure
  * Valvular disease with documented cardiac function compromise
  * Poorly controlled hypertension (i.e., diastolic BP > 100 mm Hg)

    * Patients with well-controlled hypertension and on medication are eligible for study
* Psychiatric or addictive disorders that would preclude obtaining informed consent

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Concurrent noncancer therapies allowed if used for conditions other than breast cancer
* Adjuvant therapy after surgery allowed

Exclusion criteria:

* Prior radiotherapy, chemotherapy, immunotherapy, and/or hormonal therapy for breast cancer
* Prior anthracycline therapy for any condition
* Concurrent hormonal therapy including tamoxifen, aromatase inhibitors, or raloxifene
* Concurrent sex hormonal therapy including birth-control pills or ovarian hormonal replacement therapy
* Concurrent other cancer therapy
* Concurrent herbal or alternative therapies for breast cancer

Max Age: 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey O'Connor, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel: DOXIL 30 mg/m2 + Docetaxel 60 mg/m2 every 21 days x 6 cycles Pegylated Filgrastim given on day 2 or 3 post chemotherapy
Period: Overall Study
Arm/Group | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response
Time Frame: Mammogram done pre-treatment and after four and six cycles of study chemotherapy treatment.
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel
Number analyzed (Participants) | 0

2. Primary Outcome: Clinical Complete Response
Time Frame: Surgery done after completion of six cycles of study chemotherapy treatment.
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Clinical Local Regional Response
Time Frame: Mammogram done pre-treatment and after four and six cycles of study chemotherapy treatment.
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Women Who Would Have Required a Mastectomy Upfront But Who Underwent Breast Conservation Therapy Instead After Neoadjuvant Chemotherapy
Time Frame: Baseline (pre-treatment) surgical assessment, and post-chemotherapy surgical outcome.
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel
Number analyzed (Participants) | 0

5. Secondary Outcome: Safety, in Terms of Neutropenia and Cardiac Toxicity
Time Frame: Every cycle during study treatment and 8 weeks post-treatment.
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel (N=6)
Hypersensitivity (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOXIL (Pegylated Liposomal Doxorubicin) and Docetaxel (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Lacrimation increased (Eye disorders) | 5 (5)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Stomatitis (Gastrointestinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood calcium (Investigations) | 1 (1)
Blood glucose (Investigations) | 1 (1)
Blood sodium increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (14)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Heat rash (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (5)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (5)
Flushing (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 4 (6)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and inadequate number of patients, no patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes